CLINICAL TRIAL: NCT01612221
Title: A Phase II Placebo-controlled Intervention Trial of Oral N-acetylcysteine (NAC) for Protection of Human Nevi Against UV-induced Oxidative Stress/Damage in Vivo
Brief Title: Oral N-acetylcysteine for Protection of Human Nevi Against UV-induced Oxidative Stress/Damage in Vivo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HCI50308
Record Dates: First submitted 2012-05-31; First posted 2012-06-05 (Estimated); Results first posted 2017-07-31 (Actual); Last update posted 2017-07-31 (Actual); Status verified 2017-06

CONDITIONS: Patients at Risk for Melanoma
MeSH Terms: interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patients receiving N-acetylcysteine (Experimental): Patients receiving NAC (N-acetylcysteine)
  Interventions: Drug: N-acetylcysteine
- Placebo Group (Placebo Comparator): Participants not receiving NAC (N-acetylcysteine)
  Interventions: Other: Placebo arm

INTERVENTIONS:
Drug: N-acetylcysteine — N-acetylcysteine (NAC), 1200 mg Oral route 2 doses
  Other Names: NAC
  Arms: Patients receiving N-acetylcysteine
Other: Placebo arm — Sterile normal saline, diluted into 25 cc tomato juice, orally, x 1 dose. Then repeated 24 hours later.
  Arms: Placebo Group

SUMMARY:
This is a phase II intervention to propose a new melanoma chemoprevention agent. The investigators believe oxidative stress/damage in nevi is a probable indication for melanoma risk, and propose that reduced melanoma risk in humans can be inferred by protection of nevi from ultraviolet light (UV)-induced oxidative changes. The investigators will 1) evaluate whether administration of NAC around the time of UV exposure will reduce melanoma risk in high-risk patient populations with genetic susceptibility to UV-induced oxidative stress, and 2) examine key genetic variants that will identify which individuals are most likely to benefit from chemoprotection.

ELIGIBILITY:
Inclusion Criteria:

* Must have at least 2 nevi (each >6 mm diameter) not clinically suspicious for melanoma that can be biopsied.
* Must be able to receive informed consent and sign an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria:

* The patient is a minor (< 18 years old).
* The patient cannot speak/understand English or Spanish. (NOTE: A Spanish consent form and certified interpreter can be made available if needed)
* The patient is pregnant. (NOTE: All female patients who have not had a hysterectomy and are not post-menopausal (i.e. post-menopausal for 1 year and not of child-bearing potential) will have a urine pregnancy test.)
* The patient is a prisoner, critically or mentally ill, or otherwise incapacitated or considered vulnerable.
* The patient has history of allergic reaction to NAC.
* The patient has history of severe asthma.
* The patient has been taking NAC or any other oral antioxidant.
* The patient has recent history (i.e., 3 months) of sunless tanning (tanning bed) or extensive sunburn.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-09; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Grossman, MD, PhD, Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Group: Participants not receiving NAC (N-acetylcysteine)
  Placebo arm: Sterile normal saline, diluted into 25 cc tomato juice, orally, x 1 dose.
  Then repeated 24 hours later.
Period: Overall Study
Arm/Group | Patients Receiving N-acetylcysteine | Placebo Group
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients Receiving N-acetylcysteine | Placebo Group | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 47 | 46 | 93
  >=65 years | 3 | 4 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 17 | 39
  Male | 28 | 33 | 61
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 50 | 50 | 100
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: UV-induced Oxidative Stress in Irradiated and Unirradiated Nevi
Description: Differences in the median percent nevus with 8-OG expression in UV-irradiated nevi compares with unirradiated nevi.
Time Frame: 3.5 years
Population: One subject with low-risk MC1R randomized to drug was excluded from both analyses because the lesions removed were seborrheic keratoses and not nevi, and 2 subjects (one high-risk MC1R randomized to drug and one low-risk MC1R randomized to placebo) were excluded from analysis of 8-OG because there was insufficient tissue.
Measure: Mean (Standard Deviation); unit: percentage of 8-OG expression in nevi
Arm/Group | Patients Receiving N-acetylcysteine | Placebo Group
Number analyzed (Participants) | 48 | 49
percentage of 8-OG expression in nevi
  UV Irradiated | 94.6 (12.3) | 96.2 (7.5)
  Unirradiated | 33.6 (25.1) | 33.1 (24.2)
Statistical Analysis 1: Comparison: Patients Receiving N-acetylcysteine vs Placebo Group; Test type: Superiority; p = .65, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Transcriptional Markers of UV-induced Oxidative Stress in Nevi
Description: Biomarkers susceptible to UV-induced damage protected by NAC (N-acetylcysteine) in irradiated and unirradiated nevi
Time Frame: 3.5 years
Population: One subject with low-risk MC1R randomized to drug was excluded because the lesions removed were seborrheic keratoses and not nevi.
Measure: Mean (Standard Deviation); unit: markers of UV-induced oxidative stress
Arm/Group | Patients Receiving N-acetylcysteine | Placebo Group
Number analyzed (Participants) | 49 | 50
markers of UV-induced oxidative stress
  GCLM Biomarker | 8.99 (.83) | 9.14 (.75)
  SLC1A4 Biomarker | 9.29 (.87) | 9.40 (1.06)
  SLC7A11 Biomarker | 8.73 (1.13) | 9.03 (.95)
Statistical Analysis 1: Comparison: Patients Receiving N-acetylcysteine vs Placebo Group; GCLM Biomarker analysis; Test type: Superiority; p = 0.76, ANCOVA
Statistical Analysis 2: Comparison: Patients Receiving N-acetylcysteine vs Placebo Group; SLC1A4 Biomarker analysis; Test type: Superiority; p = 0.63, ANCOVA
Statistical Analysis 3: Comparison: Patients Receiving N-acetylcysteine vs Placebo Group; SLC7A11 Biomarker analysis; Test type: Superiority; p = 0.27, ANCOVA

ADVERSE EVENTS:
Arm/Group | Patients Receiving N-acetylcysteine | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes